CLINICAL TRIAL: NCT01780103
Title: Sonographic Follow up in Newborns Diagnosed With Prenatal Hydronephrosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr Sylvia Foldi, Neonatologist MD, Hillel Yaffe Medical Center
Other Study IDs: HYMC-0055-12-CTIL
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Pyelectasis of Newborns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this retrospective study the investigators will enroll newborns that were born between 01.01.2010 and 31.12.2012 in Hillel Yaffe Medical Center with the prenatal diagnosis of Pyelectasis according to prenatal sonographic screening test.

These babies underwent renal sonography at the age of 2-5 days according to the protocol and were invited to an additional renal sonographic screening test at the age of 1 month.

The investigators will compare the results of the 2 examinations and the investigators will try to reach conclusions whether there is correspondence between the severity of the pyelectasis in the first and second sonographic tests and the outcome of these newborn babies

ELIGIBILITY:
Inclusion Criteria:

* All newborns that were born at Hillel Yaffe Medical Center with prenatal diagnosis of Hydronephrosis between 01.01.2010-31.12.2012

Exclusion Criteria:

* None

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborns at the age of 0-1 months
Sampling Method: Non-Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
severity of hydronephrosis by sonographic measures | 2 years